CLINICAL TRIAL: NCT03779399
Title: Lymphocyte T Regulatory , Th17 and NKT in Epithelial Ovarian Tumor- Prognostic Assessment and Relationship With Clinical Marker
Brief Title: Treg, Th17 Cells, NKT in Epithelial Ovarian Tumor
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Paweł Miotła, Clinical Proffesor, Medical University of Lublin
Other Study IDs: 032018
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Cancer; Borderline Ovarian Tumors; Benign Ovarian Tumor; Unexplained Infertility
Keywords: Ovarian Cancer; Borderline Ovarian Tumor; Benign Ovarian Tumor; lymphocyte T regulatory; Natural Killer T cell; ROMA; HE4
MeSH Terms: conditions — Ovarian Neoplasms | interventions — CA-125 Antigen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, ovarian tissue, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patient with benign ovarian tumor: 25 patients with benign ovarian tumor (cystadenoma) were admitted to IInd Department of Gynecology, Lublin Medical University, Lublin, Poland.
  Interventions: Other: Assessment of percentage of Treg, Th17, NKT and serum level of HE4, CA125 and ROMA.
- Patient with borderline tumor: 11 women with borderline ovarian tumor were admitted to IInd Department of Gynecology
  Interventions: Other: Assessment of percentage of Treg, Th17, NKT and serum level of HE4, CA125 and ROMA.
- Patient with ovarian cancer: 24 women with ovarian cancer were admitted to IInd Department of Gynecology
  Interventions: Other: Assessment of percentage of Treg, Th17, NKT and serum level of HE4, CA125 and ROMA.
- Patient without ovarian pathology: 20 patient with unexpleined infertility were admitted to IInd Department of Gynecology
  Interventions: Other: Assessment of percentage of Treg, Th17, NKT and serum level of HE4, CA125 and ROMA.

INTERVENTIONS:
Other: Assessment of percentage of Treg, Th17, NKT and serum level of HE4, CA125 and ROMA. — Treg, Th17, NKT cells in peripheral blood and ovarian tissue and serum level of HE4, CA125 and ROMA.

SUMMARY:
The aim of the study was to estimate the percentage and of Treg, Th17 and NKT in peripheral blood and the tissue of the epithelial ovarian tumor and relationship with blood serum level of HE4, CA125, as well as algorithm ROMA.

Material and methods Mononuclear cells (PBMCs) were isolated by density gradient centrifugation obtained from peripheral blood and ovarian tissue of patient suffering ovarian pathology. Patient from control group underwent surgery for unexplanied infertility. The percentage of Treg and Th17 , NKT in peripheral blood and the tissue was assessed using the flow cytometry method according to the manufacturer's instructions. The ROMA index was calculated according to the levels of HE4 and CA-125 in serum.

DETAILED DESCRIPTION:
Study groups. The study group consisted of 60 women. The patients were divided into 3 subgroups: a group of 24 women with malignant epithelial ovarian tumors (cystadenocarcinomas), 25 women with benign ovarian tumors (cystadenomas) and 11 women with borderline ovarian tumors (serous borderline tumors). The control group consisted of 20 women without ovarian pathology who underwent surgery for unexplanied infertility. Patients were admitted to IInd Department of Gynecology, Lublin Medical University, Lublin, Poland, between 2011 and 2014. All women with OCs were staged III or IV according to revised 2013 FIGO classification (International Journal of Gynecology and Obstetrics, January, 2014) Isolation of mononuclear cells from peripheral blood (PBMCs). Immediately after being taken from the antecubital vein, mononuclear cells (PBMCs) were isolated by density gradient centrifugation applying Gradisol L formulation of specific gravity 1.077g/ml (Aqua Medica, Łódź, Poland) for 20 min. at 700 x g. The pellet containing PBMC was washed twice in PBS and evaluated for the number (using Neubauer chamber) and viability (trypan blue staining - 0.4% trypan Blue Solution, Sigma-Aldrich, Munich, Germany). Viability of less than 95% was a disqualifying criterion.

Isolation of mononuclear cells infiltrating the tumor and healthy tissues.

During the surgery, ovarian tissue (size of approximately 1cm3) not containing any visible necrotic areas was collected. It was minced with a scalpel, suspended in 30 ml of RPMI 1640 medium (Biochrome, Holliston MA, USA) and subjected to cleavage in a mixture containing: 1 mg/ml collagenase type IA (Sigma-Aldrich, Munich, Germany), 1 mg/ml DNase type I (Sigma-Aldrich, Munich, Germany), 0.1 mg/ml hyaluronidase (Sigma-Aldrich, Munich, Germany) at 37°C for 60 min., constantly vortexed. After cleavage, the suspension was filtered through a strainer (70μm, BD Biosciences, San Jose CA, USA) and centrifuged for 5 min. at 700 x g. The suspension cells were washed twice in RPMI 1640.

Evaluation of the percentage of Th17 cells.

The evaluation of the percentage of Th17 cells (secreting IL-17A) of peripheral blood mononuclear cells, healthy tissue and tumor tissue was performed by flow cytometry using a Th17 Cytokine Staining panel according to the manufacturer's recommendation (eBiosciences, San Diego, USA) using a FACSCanto (BD Biosciences, San Jose CA,USA).

Establishment of PBMC culture and ovarian tissue (tumor or control) and stimulation with ionomycin.

After 24-hour culture of the PBMCs and ovarian tissue was set up. The medium was prepared consisting of 97% RPMI 1640 (Biochrome, Holliston MA,USA) supplemented with 2mM L-glutamine, 2% human albumin (ZLB Bioplasma, Bern, Switzerland) and antibiotics in an amount of 100 U/ml penicillin (Sigma-Aldrich, Munich, Germany) and 100 mg/ml streptomycin (Sigma-Aldrich, Munich, Germany). Cultivation was carried out in 6-well plates in a 5 ml culture medium. For each patient, two cultures were established, one of the PBMC and the other from tumor cells or normal ovarian tissue. The culture was conducted in an incubator under standard conditions (5% CO2, 95% humidity, 37°C) for 4 hours. To individual wells were added: ionomycin (Sigma-Aldrich, Munich, Germany) at a concentration of 1 ug/ml and PMA at a concentration of 25 ng/ml to stimulate cells for the production of cytokines and brefeldin at a concentration 10 μg/ml (Sigma-Aldrich, Munich, Germany) in order to inhibit the activity of the endoplasmic reticulum, leading to retain the cytokine within the cell.

The determination of intracellular cytokines.

24-hour cultures after moving from the culture plate to two properly signed tubes were washed twice in 2 ml of Flow Cytometry Staining Buffer (eBioscience, San Diego, USA) after vortexing. Constant parameters used during each rinsing in this procedure are: run time 5 min., 700 x g. After removing the supernatant, 5μl of anti-CD4 (eFluor 450, eBioscience, San Diego, USA) was added to each tube. The mixture was incubated for 20 min. in darkness. After washing away, the excess of antibody in 2 ml of Flow Cytometry Staining Buffer (eBioscience, San Diego,USA), 100μl IC Fixation Buffer (eBioscience, San Diego, USA) was added to each tube in order to consolidate. Mixing/Vortexing this mixture was also incubated for 20 minutes in darkness. Then it was washed twice with 2 ml of the permeabilization buffer (Permeabilization Buffer, eBioscience, San Diego, USA). Preparing the buffer involved its 10-fold dilution with PBS. After removing the supernatant, the cells were resuspended in 100μl of permeabilization buffer and separated to previously prepared cytometry tubes into control and test samples. Thereafter, 5μl antibodies were added to the test samples: anti-IL-17A (FITC). After vortexing, all samples were incubated for 20 min. in darkness. They were washed twice and after suspending the cells in the Flow Cytometry Staining Buffer, cytometric analysis was carried out. Analysis was performed using flow cytometric BD FACSCanto II (BD Biosciences, San Diego, USA). Measurements were performed using the software BDFACS Diva.

Estimation of the percentage of regulatory T lymphocytes.

Estimation of the percentage of regulatory T lymphocytes among peripheral blood mononuclear cells and in healthy and neoplastic tissue was made with the flow cytometry method using the Human Treg Flow™ Kit (FOXP3 Alexa Fluor® 488 / CD4 PE-Cy5/CD25 PE, BioLegend®, USA) with the use of FACSCanto apparatus (BD Biosciences, San Diego,USA).

Determination of iNKT cell subpopulation by flow cytometry

Mononuclear cells isolated from peripheral blood, healthy tissue and epithelial ovarian tumors were incubated with the appropriate volume (according to the procedures recommended by the manufacturers) of the appropriate monoclonal antibodies: the anti-iNKT FITC (anti-Vα24) (cat#558371, clone 6B11, BD Pharmingen, San Jose, CA, USA), anti-CD3 PE (Cat #554829, clone G4. 18, BD Pharmingen, San Jose, CA, USA) and anti CD161-PE f(clone Dx12, Cat#550968, BD Pharmingen, San Jose, CA, USA). Prepared samples were incubated for 20 min. at room temperature in the dark. After twice washing in buffered physiological saline (PBS), the cells were immediately subjected to cytometric analysis. Data acquisition and analysis were performed using a FACS Calibur flow cytometer (Becton Dickinson, New Jersey, USA). Expressing cells iNKT+/CD3+/CD161+ were rated among CD3+

Assessment of concentration of protein HE4, CA125 and algorithm ROMA.

Samples were collected from all the patients prior to surgery and 3 ml blood was collected. Serum was centrifuged at 2000 × g and stored at -20 and -80°C until use. Serum level of CA-125 and HE4 were detected using the full automatic chemiluminescence analyzer Cobs601 and the test procedure was performed according to the manufacturer's instructions (Roche Diagnostics, Indianapolis, IN, USA). Next, serum HE4 and CA-125 levels were calculated for ROMA index value using the Roche ROMA index of ovarian cancer risk assessment software. Serum HE4 and CA-125 reference range was <140 pmol/l and <32 U/ml, respectively.

Assessment of risk of epithelial ovarian carcinoma (ROMA) The ROMA index was calculated according to the levels of HE4 and CA-125. HE4 and CA-125 amount were input to the ovarian cancer risk assessment software, followed by automatic calculation of the corresponding ROMA index. The premenopausal calculation formula of the ROMA index was: 12+2.38 × LN(HE4)+0.062 6 × LN(CA-125). The postmenopausal calculation formula of the ROMA index was: 8.09+1.04 × LN(HE4)+0.732 × LN(CA-125). Premenopausal women with a ROMA value ≥11.4, had a higher risk of ovarian cancer. Postmenopausal women with ROMA value ≥29.9 had a higher risk of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age 18-75
* ovarian tumor

Exclusion Criteria:

* below 18 years old
* necrosis in tumor

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75
Study Population: The study group consisted of 60 women. The patients were divided into 3 subgroups: a group of 24 women with malignant epithelial ovarian tumors (cystadenocarcinomas), 25 women with benign ovarian tumors (cystadenomas) and 11 women with borderline ovarian tumors (serous borderline tumors). The control group consisted of 20 women without ovarian pathology who underwent surgery for unexplanied infertility. Patients were admitted to IInd Department of Gynecology, Lublin Medical University, Lublin, Poland, between 2011 and 2014. All women with OCs were staged III or IV according to revised 2013 FIGO classification (International Journal of Gynecology and Obstetrics, January, 2014)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Treg, Th17, NKT in peripheral blood and tissue | 3 days
  Percentage of regulatory TREG, Th17, NKT among peripheral blood mononuclear cells and in healthy and neoplastic tissue was made with the flow cytometry
Value of ROMA in serum | 3 days
  Assessment level of CA125 and HE4 in serum

SECONDARY OUTCOMES:
Prognostic assessment of T reg, Th17, NKT lymphocytes in the tissue and peripheral blood of patients with ovarian cancer | 3 years
  Kaplan-Meier survival analysis was performed in the group of patients with ovarian cancer.
Association between Treg, Th17,NKTand clinical marker | 1 year
  Spearman's rank correlation coefficient and its significance test was applied to assess relationships between two parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Izabela Winkler, Principal Investigator — Medical University of Lublin
Locations (1):
- IInd Department of Gynecology, Lublin, Poland

REFERENCES:
- [Derived] Winkler I, Wos J, Bojarska-Junak A, Semczuk A, Rechberger T, Baranowski W, Markut-Miotla E, Tabarkiewicz J, Wolinska E, Skrzypczak M. An association of iNKT+/CD3+/CD161+ lymphocytes in ovarian cancer tissue with CA125 serum concentration. Immunobiology. 2020 Nov;225(6):152010. doi: 10.1016/j.imbio.2020.152010. Epub 2020 Aug 28. PMID 33130518